CLINICAL TRIAL: NCT03819114
Title: An Open-Label, Phase II Pharmacokinetic Study to Evaluate Double-Dose Levonorgestrel Emergency Contraception in Combination With Efavirenz-Based Antiretroviral Therapy or Rifampicin-Containing Anti-Tuberculosis Therapy
Brief Title: Pharmacokinetic Study to Evaluate Double-Dose Levonorgestrel Emergency Contraception in Combination With Efavirenz-Based Antiretroviral Therapy or Rifampicin-Containing Anti-Tuberculosis Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5375; 38493 (Registry Identifier: DAIDS-ES Registry Number); UM1AI068636 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Levonorgestrel; Pharmacokinetics; Efavirenz; Dolutegravir; Rifampin
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A: LNG 1.5 mg among participants on EFV-based ART (randomized) (Experimental): Participants received 1.5 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
  Interventions: Drug: Levonorgestrel (LNG)
- B: LNG 3.0 mg among participants on EFV-based ART (randomized) (Experimental): Participants received 3mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
  Interventions: Drug: Levonorgestrel (LNG)
- C: LNG 1.5 mg among participants on DTG-based ART (assigned) (Experimental): Participants received 1.5 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
  Interventions: Drug: Levonorgestrel (LNG)
- D: LNG 3.0 mg among participants on RIF-INH TB Therapy (assigned) (Experimental): Participants received 3mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
  Interventions: Drug: Levonorgestrel (LNG)

INTERVENTIONS:
Drug: Levonorgestrel (LNG) — LNG tablet(s) were administered by mouth in a directly observed manner.

SUMMARY:
The purpose of this pharmacokinetic (PK) study was to evaluate if a double dose (3 mg) of levonorgestrel (LNG) overcomes known drug-drug interactions (DDIs) with efavirenz (EFV)-based antiretroviral therapy (ART) or rifampicin (RIF)-containing tuberculosis (TB) therapy. The safety of double-dose (3.0 mg) LNG versus standard-dose (1.5 mg) was also compared.

DETAILED DESCRIPTION:
This pharmacokinetic (PK) study evaluated if a double dose (3.0 mg) of levonorgestrel (LNG) overcomes known drug-drug interactions (DDIs) with efavirenz (EFV)-based antiretroviral therapy (ART) or rifampicin (RIF)-containing tuberculosis (TB) therapy. The safety of double-dose (3.0 mg) LNG versus standard-dose (1.5 mg) was also compared.

Participants were volunteers who did not require emergency contraception (EC) for contraception at the time of trial participation. This trial enrolled persons assigned female sex at birth who were 16 years of age or older. Group assignment was determined by disease status (HIV or TB; participants could not have been living with both HIV and TB), and, for those with HIV, by ART regimen at enrollment. Participants with HIV who were taking EFV-based ART were randomized to receive a standard dose LNG (Group A) or a double dose of LNG (Group B). Participants taking dolutegravir (DTG)-based ART were assigned to a standard dose of LNG (Group C). Participants in the continuation phase of active TB treatment taking RIF and isoniazid (INH) with or without ethambutol were assigned to a double dose of LNG (Group D).

At study entry, participants in Groups A and C received a standard single dose of LNG. Participants in Groups B and D received a double dose of LNG. Intensive PK monitoring was conducted pre-dose, and after the LNG dose. Participants were expected to remain at the clinical site while the initial 8 hour PK samples were collected, and to return to the clinical site for the 24 and 48 hour samples.

All participants completed self-report questionnaires to assess adherence to TB therapy and ART, menstrual history and patterns after LNG administration, and to collect adverse effects commonly reported with LNG (i.e., irregular bleeding patterns). Adherence to ART and RIF was also assessed by collecting hair samples and single plasma concentrations at entry. Participants were followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenarcheal female.

  * Note: Participant report and clinician's opinion were acceptable.
* The following laboratory values obtained within 30 days prior to study entry by any US laboratory that had a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any ACTG network-approved non-US laboratory that operated in accordance with Good Clinical Laboratory Practices (GCLP) and participated in appropriate external quality assurance (EQA) programs.

  * Absolute neutrophil count (ANC) greater than or equal to 500 cells/mm^3
  * Platelet count greater than or equal to 50,000 platelets/mm^3
  * Hemoglobin greater than or equal to 8.0 g/dL
  * Aspartate transaminase (AST) less than 5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) less than 5 x ULN
  * Creatinine less than or equal to 1.5 x ULN
  * Total bilirubin less than or equal to 2.0 x ULN
* Negative serum or urine pregnancy test within 30 days prior to study entry and within 48 hours prior to entry (if screening occurred more than 48 hours prior to entry) by any US clinic or US laboratory that had a CLIA certification or its equivalent, or used a point of care (POC)/CLIA-waived test, or at any network-approved non-US laboratory or non-US clinic that operated in accordance with GCLP and participated in appropriate EQA programs. The serum or urine pregnancy test must have had a sensitivity of at least 25 mIU/mL.
* Had not had sex that could lead to pregnancy without contraception within 14 days prior to study entry as defined in the criteria below, according to participant self-report.
* Contraception requirements

  * All participants agreed not to participate in a conception process (e.g., active attempt to become pregnant or in vitro fertilization) for the duration of the study. Women of reproductive potential, who were participating in sexual activity that could lead to pregnancy, agreed to use at least one reliable method of contraception while in the study. Acceptable forms of contraceptives included:

    * Male condom with or without a spermicidal agent
    * Diaphragm or cervical cap with spermicide
    * Non-hormonal intrauterine device (IUD)
    * Bilateral tubal ligation
    * Male partner vasectomy
* Ability and willingness of participant or legal guardian/representative to have provided informed consent.
* Body mass index (BMI) (kg/m^2) available at entry. See the study protocol for BMI calculation instructions.

  * Note: A maximum of 5 participants with BMI greater than or equal to 30 kg/m^2 were allowed in each arm B-D and a maximum of 3 participants in Arm A.
* For participants with HIV: HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

  * Note: The term "licensed" referred to a US Food and Drug Administration (FDA)-approved kit, which was required for all investigational new drug (IND) studies, or for sites located in countries other than the United States, a kit that had been certified or licensed by an oversight body within that country and validated internally. Non-US sites were encouraged to use US FDA-approved methods for IND studies.
  * World Health Organization (WHO) and Centers for Disease Control and Prevention (CDC) guidelines mandated that confirmation of the initial test result must have used a test that was different from the one used for the initial assessment. A reactive initial rapid test was confirmed by either another type of rapid assay or an E/CIA that was based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* For participants with HIV: Received a stable qualifying concomitant ART regimen containing either once-daily DTG 50 mg or EFV 600 mg with no changes in the components of their ART for at least 30 days prior to study entry.
* For participants who were being treated for TB: HIV-negative at screening, documented within the prior 6 months by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, or plasma HIV-1 RNA viral load.

  * Note: The term "licensed" referred to a US FDA-approved kit, which was required for all IND studies, or for sites located in countries other than the United States, a kit that had been certified or licensed by an oversight body within that country and validated internally. Non-US sites were encouraged to use US FDA-approved methods for IND studies.
  * WHO and CDC guidelines mandated that confirmation of the initial test result must have used a test that was different from the one used for the initial assessment. A reactive initial rapid test was confirmed by either another type of rapid assay or an E/CIA that was based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* For participants who were living without HIV and being treated for TB: Received RIF and INH on a once daily dosing (7 days per week) schedule at study entry, after completion of the intensive phase of TB treatment.

  * Note: Inclusion of ethambutol as part of continuation phase of TB therapy was allowed.
* Ability and willingness of participant to have been contacted remotely for study visits.

Exclusion Criteria

* Known allergy/sensitivity or any hypersensitivity to LNG or components of the formulation.
* Bilateral oophorectomy, hysterectomy, or postmenopausal

  * Note: Postmenopausal was defined as amenorrhea for at least 12 consecutive months prior to study entry (in the absence of medications known to induce amenorrhea), and had a documented follicle stimulated hormone-release factor (FSH) measurement greater than 40 mIU/mL or a result in the testing laboratory's menopausal range. If an FSH level was not available, 24 consecutive months of amenorrhea prior to study entry (in the absence of medications known to induce amenorrhea).
  * Note: Clinical assessment and clinician's opinion were acceptable.
* Was currently pregnant, was within 6 weeks of delivery, or was currently breastfeeding an infant under 6 months of age.

  * Note: For recent pregnancy resolution during the first or second trimester, the participant was only eligible when the pregnancy test result was negative.
* Receipt of LNG within 30 days prior to study entry.
* Receipt of depo-medroxyprogesterone for 90 days prior to study entry, or norethisterone enanthate (NET-EN) within 60 days prior to study entry, or other hormonal contraceptives within 30 days prior to study entry.
* Used any drugs other than RIF and EFV known to: 1) induce CYP3A4 system within 30 days prior to study entry, and 2) inhibit the CYP3A4 system within 7 days prior to study entry. See the study protocol for prohibited and precautionary medications.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would have interfered with adherence to study requirements.
* Acute or serious illness that required systemic treatment and/or hospitalization within 14 days prior to study entry.
* Other medical, psychiatric, or psychological condition that, in the opinion of the site investigator, would have interfered with completion of study procedures and or adherence to study drug.
* For participants with HIV: Was currently receiving medications for TB infection.
* For participants with HIV: Had missed one or more of the prescribed doses of HIV medications within 3 days prior to study entry.

  * Note: The entry visit could have been rescheduled within the screening period once the participant had taken all prescribed doses within 3 days prior to study entry.
* For participants who were not living with HIV and were being treated for TB: Had missed one or more of the prescribed doses of TB medication within 3 days prior to study entry.

  * Note: The entry visit could have been rescheduled within the screening period once the participant had taken all prescribed doses within 3 days prior to study entry.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Scarsi, PharmD, MS, Study Chair — Northwestern University CRS, University of Nebraska Medical Center
Locations (18):
- United States (7):
  - 2701 Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Weill Cornell Upton CRS (7803), New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pitt CRS (1001), Pittsburgh, Pennsylvania
  - Trinity Health and Wellness Center CRS (31443), Dallas, Texas
- Gaborone CRS (12701), Gaborone, Botswana
- 12101 Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS (12501), Kericho, Kenya
- Malawi (2):
  - Blantyre CRS (30301), Blantyre
  - Malawi CRS (12001), Lilongwe
- South Africa (4):
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (11101), Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CUR) CRS (8950), Cape Town, West Cape
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
- Thailand (2):
  - 31802 Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok, Patumwan
  - 31784 Chiang Mai University HIV Treatment CRS, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.1, July 2017. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: DAIDS AE Grading Table Addendum 1, Female Genital Grading Table for Use in Microbicide Studies, Version 1.0, November 2007 — https://rsc.niaid.nih.gov/sites/default/files/addendum-1-female-genital-grading-table-v1-nov-2007.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from 18 sites. Sites were located in the United States and internationally (Botswana, Brazil, Kenya, Malawi, South Africa, Thailand). The first participant accrued in May 2019, and the last participant accrued in November 2020.
Pre-assignment Details: Participants receiving EFV-based ART therapy were randomized between Group A (1.5mg dose of LNG) and Group B (3.0mg dose of LNG) in a 1:2 ratio using permuted blocks and institutional balancing. Participants living with HIV receiving DTG-based ART therapy and participants with TB receiving RIF-INH therapy were assigned to study groups C and D, respectively.
  Women with BMI greater than or equal to 30 kg/m2 were limited to no more than 5 within Groups B-D and no more than three within Group A.
Groups:
- B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned): Participants received 3 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
Period: Overall Study
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Started | 17 | 36 | 35 | 34
Received LNG Treatment | 17 | 36 | 35 | 34
Completed | 17 | 35 | 33 | 34
Not Completed | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who took assigned dose of LNG and prescribed doses of background drugs (ART or TB treatment) and who had LNG PK concentrations available over the sampling time frame.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned) | Total
Number analyzed (Participants) | 17 | 35 | 32 | 34 | 118
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [35 to 45] | 36 [29 to 42] | 34 [29 to 40] | 25 [21 to 35] | 34 [27 to 41]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 17 | 35 | 32 | 34 | 118
    Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 20 | 2 | 2 | 33
  Black (Non-Hispanic) | 7 | 12 | 24 | 30 | 73
  Hispanic or Latino (Regardless of race) | 1 | 3 | 4 | 2 | 10
  Multiple Races | 0 | 0 | 1 | 0 | 1
  White (Non-Hispanic) | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Botswana | 0 | 0 | 0 | 2 | 2
  Brazil | 1 | 3 | 4 | 2 | 10
  Kenya | 0 | 0 | 0 | 4 | 4
  Malawi | 0 | 0 | 10 | 6 | 16
  South Africa | 7 | 12 | 2 | 18 | 39
  Thailand | 9 | 20 | 2 | 2 | 33
  United States | 0 | 0 | 14 | 0 | 14
Gender Identity [Count of Participants; unit: Participants]
  Cisgender | 17 | 35 | 32 | 34 | 118
  Transgender spectrum | 0 | 0 | 0 | 0 | 0
HIV-1 Infection Status [Count of Participants; unit: Participants]
  HIV-1 infection present | 17 | 35 | 32 | 0 | 84
  HIV-1 infection absent | 0 | 0 | 0 | 34 | 34

OUTCOME MEASURES:

1. Primary Outcome: LNG Area Under the Concentration-time Curve (AUC0-8h) Calculated Based on Intensive LNG PK Samples Obtained From Individual Participants
Description: AUC for each participant was calculated from all available LNG concentrations measured over 8 hours using the linear up/log down version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule used linear interpolation between untransformed data up to Cmax, and between log-transformed data from Cmax through Clast. Assay lower limit of quantification (LLOQ) for LNG was 0.025 ng/mL; values < LLOQ were imputed as 0 (if pre-dose) or as 0.0125 (if post-dose).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours * ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours * ng/mL | 52.13 [36.72 to 88.27] | 102.13 [64.52 to 114.75] | 80.50 [66.64 to 125.06] | 124.39 [87.10 to 168.79]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Equivalence — Confidence Interval (CI) on Geometric Mean Ratio compared to reference interval (0.7, 1.43); Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.81 to 1.20] — The ratios of the geometric means (group B / group C) and its 90% CI were obtained by exponentiating the least squares mean difference and its 90% CI of the natural log-transformed data
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Equivalence — Confidence Interval on Geometric Mean Ratio compared to reference interval (0.7, 1.43); Geometric Mean Ratio = 1.34, 90% CI 2-sided [1.12 to 1.60] — The ratios of the geometric means (group D / group C) and its 90% CI were obtained by exponentiating the least squares mean difference and its 90% CI of the natural log-transformed data
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Superiority — Confidence Interval on Geometric Mean Ratio excluding 1; Geometric Mean Ratio = 1.66, 90% CI 2-sided [1.27 to 2.18] — The ratios of the geometric means (group B / group A) and its 90% CI were obtained by exponentiating the least squares mean difference and its 90% CI of the natural log-transformed data
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Superiority — Confidence Interval on Geometric Mean Ratio excluding 1; Geometric Mean Ratio = 0.59, 90% CI 2-sided [0.45 to 0.78] — The ratios of the geometric means (group A / group C) and its 90% CI were obtained by exponentiating the least squares mean difference and its 90% CI of the natural log-transformed data

2. Secondary Outcome: Number and Percentage of Participants Experiencing Either a Serious Adverse Event (SAE) or Adverse Event (AE) Potentially or Definitely Associated With Single Dose LNG Administration.
Description: Adverse events were Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 and DAIDS AE Grading Table Addendum 1, Female Genital Grading Table for Use in Microbicide Studies, Version 1.0 - November 2007. Relationship of AE to study treatment was determined by the site, study core team, and DAIDS clinical representative.
  AEs evaluated in this outcome fulfilled the below criteria:
  * Potentially or definitely related to LNG dose
  * Grade 3 or higher AEs
  * Grade 2 of higher nausea, diarrhea, menorrhagia or metrorrhagia, and ectopic pregnancies
Time Frame: From Day 0 through study Day 28
Population: Participants who received LNG study treatment, grouped by LNG dose. LNG 1.5mg includes Group A (LNG 1.5 mg Among Participants on EFV-based ART (Randomized)) and Group C (LNG 1.5 mg Among Participants on DTG-based ART (Assigned)) participants. LNG 3.0mg includes Group B (LNG 3.0 mg Among Participants on EFV-based ART (Randomized)) and Group D (LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)) participants.
Measure: Count of Participants; unit: Participants
Groups:
- LNG 1.5 mg: Participants received 1.5 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
- LNG 3.0 mg: Participants received 3 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
Arm/Group | LNG 1.5 mg | LNG 3.0 mg
Number analyzed (Participants) | 52 | 70
Participants | 2 | 2
Statistical Analysis 1: Comparison: LNG 1.5 mg vs LNG 3.0 mg; Test type: Superiority; p = 1.00, Fisher Exact — No adjustments for multiple comparisons were made. Statistical significance was declared if p<0.05

3. Secondary Outcome: Maximum Concentration (Cmax) of LNG
Description: Cmax for each participant was calculated as the maximum observed LNG concentration from LNG PK samples at pre-dose through 48 hours post-dose. Standard noncompartmental techniques were used to determine Cmax using the software package Phoenix WinNonLin (Certara®).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
ng/mL | 15.10 [11.20 to 24.00] | 24.90 [16.20 to 29.60] | 18.65 [14.05 to 26.15] | 28.01 [23.00 to 39.60]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.17, 90% CI 2-sided [0.96 to 1.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.43, 90% CI 2-sided [1.21 to 1.69] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.51, 90% CI 2-sided [1.17 to 1.96] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.77, 90% CI 2-sided [0.60 to 1.00] — [estimate comment as in outcome 1, analysis 4]

4. Secondary Outcome: Minimum Concentration (Cmin) of LNG
Description: Cmin for each participant was calculated as the minimum observed LNG concentration from LNG PK samples at pre-dose through 48 hours post-dose. Standard noncompartmental techniques were used to determine Cmin using the software package Phoenix WinNonLin (Certara®). Assay lower limit of quantification for LNG was 0.025 ng/mL; values < LLOQ were imputed as 0 (if pre-dose) or as 0.0125 (if post-dose).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
ng/mL | 0.25 [0.13 to 0.37] | 0.56 [0.19 to 1.08] | 1.49 [0.80 to 3.07] | 0.41 [0.17 to 0.74]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.37, 90% CI 2-sided [0.22 to 0.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.25, 90% CI 2-sided [0.15 to 0.44] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 2.11, 90% CI 2-sided [1.20 to 3.70] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.17, 90% CI 2-sided [0.09 to 0.32] — [estimate comment as in outcome 1, analysis 4]

5. Secondary Outcome: Oral Clearance (CL/F) of LNG
Description: Apparent oral clearance (CL/F) for each participant was calculated as CL/F = dose/AUC0-24 or CL/F = dose/AUC0-48 of the observed LNG concentration from LNG PK samples at pre-dose through 48 hours post-dose. Standard noncompartmental techniques were used to determine CL/F using the software package Phoenix WinNonLin (Certara®).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: L/h
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
L/h | 12.64 [10.44 to 21.06] | 15.24 [12.59 to 27.66] | 4.39 [2.89 to 6.59] | 12.05 [9.01 to 16.32]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 4.03, 90% CI 2-sided [3.17 to 5.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 2.92, 90% CI 2-sided [2.33 to 3.65] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.11, 90% CI 2-sided [0.82 to 1.52] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 3.62, 90% CI 2-sided [2.65 to 4.93] — [estimate comment as in outcome 1, analysis 4]

6. Secondary Outcome: Volume of Distribution (Vd) of LNG
Description: Vd for each participant was calculated from observed LNG concentration from LNG PK samples at pre-dose through 48 hours post-dose. Standard noncompartmental techniques were used to determine Vd using the software package Phoenix WinNonLin (Certara®).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: L
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
L | 276.70 [118.28 to 411.82] | 294.92 [208.70 to 489.52] | 169.05 [93.83 to 215.16] | 156.31 [105.26 to 247.20]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 2.10, 90% CI 2-sided [1.66 to 2.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.11, 90% CI 2-sided [0.89 to 1.39] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.20, 90% CI 2-sided [0.87 to 1.66] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.75, 90% CI 2-sided [1.24 to 2.45] — [estimate comment as in outcome 1, analysis 4]

7. Secondary Outcome: Half-life (T1/2) of LNG
Description: T1/2 for each participant was calculated using regression analysis when possible from the observed LNG concentration from LNG PK samples at pre-dose through 48 hours post-dose. Standard noncompartmental techniques were used to determine T1/2 using the software package Phoenix WinNonLin (Certara®).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours | 12.05 [8.63 to 13.70] | 11.79 [10.58 to 13.80] | 24.03 [19.95 to 28.03] | 8.97 [6.72 to 11.89]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.52, 90% CI 2-sided [0.46 to 0.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.38, 90% CI 2-sided [0.34 to 0.43] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.08, 90% CI 2-sided [0.93 to 1.25] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.48, 90% CI 2-sided [0.41 to 0.56] — [estimate comment as in outcome 1, analysis 4]

8. Secondary Outcome: Time of Minimum Concentration (Tmin) of LNG
Description: Tmin for each participant was time to the minimum observed LNG concentration after the observed dose.
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours pose-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours | 47.07 [46.13 to 48.00] | 47.95 [46.13 to 48.00] | 47.61 [0.50 to 48.31] | 48.00 [46.55 to 48.00]

9. Secondary Outcome: LNG Area Under the Concentration Time Curve (AUC0-24h) Calculated Based on Intensive LNG PK Samples Obtained From Individual Participants
Description: AUC for each participant was calculated from all available LNG concentrations measured over 24 hours using the linear up/log down version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule used linear interpolation between untransformed data up to Cmax, and between log-transformed data from Cmax through Clast. Assay lower limit of quantification for LNG was 0.025 ng/mL; values < LLOQ were imputed as 0 (if pre-dose) or as 0.0125 (if post-dose).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours * ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours * ng/mL | 81.64 [56.14 to 128.49] | 153.40 [100.13 to 190.48] | 157.56 [132.30 to 282.32] | 213.69 [148.64 to 283.22]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.75, 90% CI 2-sided [0.60 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.10, 90% CI 2-sided [0.90 to 1.36] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.74, 90% CI 2-sided [1.29 to 2.33] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.43, 90% CI 2-sided [0.32 to 0.58] — [estimate comment as in outcome 1, analysis 4]

10. Secondary Outcome: LNG Area Under the Concentration Time Curve (AUC0-48h) Calculated Based on Intensive LNG PK Samples Obtained From Individual Participants
Description: AUC for each participant was calculated from all available LNG concentrations measured over 48 hours using the linear up/log down version of the trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule used linear interpolation between untransformed data up to Cmax, and between log-transformed data from Cmax through Clast. Assay lower limit of quantification for LNG was 0.025 ng/mL; values < LLOQ were imputed as 0 (if pre-dose) or as 0.0125 (if post-dose).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours pose-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours * ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours * ng/mL | 98.95 [66.38 to 141.27] | 180.25 [106.87 to 216.75] | 224.81 [178.30 to 400.90] | 242.68 [181.56 to 321.98]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.62, 90% CI 2-sided [0.49 to 0.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.89, 90% CI 2-sided [0.71 to 1.10] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.77, 90% CI 2-sided [1.31 to 2.40] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.35, 90% CI 2-sided [0.26 to 0.47] — [estimate comment as in outcome 1, analysis 4]

11. Secondary Outcome: LNG Total Area Under the Concentration Time Curve AUCinf (Infinity) Calculated Based on Intensive LNG PK Samples Obtained From Individual Participants
Description: AUC for each participant was calculated from all available LNG concentrations measured to infinity hours using the linear up/log down version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule used linear interpolation between untransformed data up to Cmax, and between log-transformed data from Cmax through Clast. Assay lower limit of quantification for LNG was 0.025 ng/mL; values < LLOQ were imputed as 0 (if pre-dose) or as 0.0125 (if post-dose).
Time Frame: Intensive LNG PK samples at pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours pose-dose
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours * ng/mL
Arm/Group | A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned)
Number analyzed (Participants) | 17 | 35 | 32 | 34
hours * ng/mL | 118.71 [71.23 to 143.69] | 196.83 [108.48 to 238.24] | 345.80 [227.80 to 518.69] | 248.96 [183.87 to 333.05]
Statistical Analysis 1: Comparison: B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.50, 90% CI 2-sided [0.39 to 0.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned) vs D: LNG 3.0 mg Among Participants on RIF-INH TB Therapy (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.69, 90% CI 2-sided [0.55 to 0.86] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs B: LNG 3.0 mg Among Participants on EFV-based ART (Randomized); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 1.80, 90% CI 2-sided [1.32 to 2.45] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: A: LNG 1.5 mg Among Participants on EFV-based ART (Randomized) vs C: LNG 1.5 mg Among Participants on DTG-based ART (Assigned); Test type: Other — No hypothesis testing was performed; Geometric Mean Ratio = 0.28, 90% CI 2-sided [0.20 to 0.38] — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Day 28 or premature study discontinuation.
Description: The DAIDS AE Grading Table (V2.1) and Addendum 1, Female Genital Grading Table for Use in Microbicide Studies, Version 1.0 - November 2007 were used.
  AEs were recorded on the case report forms (CRFs) if any of the following criteria had been met:
  * All Grade ≥3 AEs considered potentially or definitely related to LNG
  * All Grade ≥2 nausea, diarrhea, menorrhagia, or metrorrhagia
  * Ectopic pregnancy
  * All AEs meeting Serious Adverse Event (SAE) definition
Groups:
- A: LNG 1.5 mg Among Women on EFV-based ART (Randomized); C: LNG 1.5 mg Among Women on DTG-based ART (Assigned): Participants received 1.5 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
- B: LNG 3.0 mg Among Women on EFV-based ART (Randomized); D: LNG 3.0 mg Among Women on RIF-INH TB Therapy (Assigned): Participants received 3 mg of LNG once orally on Day 0 and were followed post-treatment for 4 weeks.
Arm/Group | A: LNG 1.5 mg Among Women on EFV-based ART (Randomized) | B: LNG 3.0 mg Among Women on EFV-based ART (Randomized) | C: LNG 1.5 mg Among Women on DTG-based ART (Assigned) | D: LNG 3.0 mg Among Women on RIF-INH TB Therapy (Assigned)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/36 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/36 | 0/35 | 1/34
Other Adverse Events (participants affected / at risk) | 1/17 | 0/36 | 1/35 | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: LNG 1.5 mg Among Women on EFV-based ART (Randomized) (N=17) | B: LNG 3.0 mg Among Women on EFV-based ART (Randomized) (N=36) | C: LNG 1.5 mg Among Women on DTG-based ART (Assigned) (N=35) | D: LNG 3.0 mg Among Women on RIF-INH TB Therapy (Assigned) (N=34)
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: LNG 1.5 mg Among Women on EFV-based ART (Randomized) (N=17) | B: LNG 3.0 mg Among Women on EFV-based ART (Randomized) (N=36) | C: LNG 1.5 mg Among Women on DTG-based ART (Assigned) (N=35) | D: LNG 3.0 mg Among Women on RIF-INH TB Therapy (Assigned) (N=34)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menstrual discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03819114/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT03819114/SAP_001.pdf
  • Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT03819114/ICF_002.pdf